CLINICAL TRIAL: NCT01121224
Title: CSP #571 - Drug-eluting Stents vs. Bare Metal Stents in Saphenous Vein Graft Angioplasty (DIVA)
Brief Title: Drug-Eluting Stents vs. Bare Metal Stents In Saphenous Vein Graft Angioplasty
Acronym: DIVA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 571
Record Dates: First submitted 2010-05-07; First posted 2010-05-12 (Estimated); Results first posted 2018-02-01 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Saphenous Vein Graft Atherosclerosis
Keywords: Saphenous vein graft; Percutaneous coronary intervention; Stents
MeSH Terms: interventions — Drug-Eluting Stents; Clopidogrel; thienopyridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- BMS Group (Active Comparator): Patients who receive a bare metal stent in the saphenous vein graft target lesion(s).
  Interventions: Device: Bare Metal Stent; Drug: Placebo; Drug: Thienopyridine (open-label)
- DES Group (Experimental): Patients who receive a drug-eluting stent in the saphenous vein graft target lesion(s).
  Interventions: Device: Drug-Eluting Stent; Drug: Blinded clopidogrel; Drug: Thienopyridine (open-label)

INTERVENTIONS:
Device: Bare Metal Stent — Patients receive one or more bare metal stents in the saphenous vein graft target lesion.
  Other Names: BMS
  Arms: BMS Group
Device: Drug-Eluting Stent — Patients receive one or more drug-eluting stents in the saphenous vein graft target lesion.
  Other Names: DES
  Arms: DES Group
Drug: Blinded clopidogrel — For non-ACS patients with no other clinical indication for open-label thienopyridine who receive one or more DES in the target lesion.
  Other Names: Plavix
  Arms: DES Group
Drug: Placebo — For non-ACS patients with no other clinical indication for open-label thienopyridine who receive only BMS.
  Arms: BMS Group
Drug: Thienopyridine (open-label) — For ACS patients who receive BMS or DES in their saphenous vein graft or patients for whom there is another clinical indication for open-label thienopyridine. Also for patients who receive a DES in a non-target lesion.

SUMMARY:
Patients who have undergone coronary bypass surgery have had a vein removed from the leg and implanted in the chest to "bypass" blockages in the coronary arteries. These veins are called saphenous vein grafts or SVGs. SVGs often develop blockages that can cause chest pain and heart attacks. SVG blockages can be opened by using small balloons and stents (metal coils that keep the artery open). Two types of stents are currently used: bare metal stents (BMS) and drug-eluting stents (DES). Both BMS and DES are made of metal. DES are also coated with a drug that releases into the wall of the blood vessel to prevent scar tissue from forming and re-narrowing the vessel. Both stents have advantages and disadvantages: DES require taking special blood thinners (called thienopyridines, such as clopidogrel or prasugrel) longer than bare metal stent and could have more bleeding but are also less likely to renarrow. Both BMS and DES are routinely being used in SVGs, but it is not known which one is better. Neither bare metal (except for an outdated model) nor drug-eluting stents are FDA approved for use in SVGs. The purpose of CSP#571 is to compare the outcomes after DES vs. BMS use in SVGs.

In CSP#571 patients who need stenting of SVG blockages will be randomized to receive DES or BMS in a 1:1 ratio. Per standard practice, patients will receive 12 months of an open label thienopyridine if they have acute coronary syndrome (ACS), or if they have another clinical reason for needing the medication. Patients without ACS who receive DES also need to take 12 months of a thienopyridine whether or not they are in the study, but non-ACS patients who receive a BMS do not. In order to make sure patients do not know which stent they received, non-ACS patients who received BMS will receive 1 month of open label thienopyridine followed by 11 months of blinded placebo, while those who received DES will receive 1 month of open label thienopyridine followed by 11 months of blinded clopidogrel, which is a thienopyridine.

All study patients will be followed in the clinic for at least 1 year after their stenting procedure to see if there is a difference in the rate of cardiac death, heart attack, or any procedure that is required in order to increase the flow of blood to and from the heart between the BMS and DES groups.

DETAILED DESCRIPTION:
VA Cooperative Studies Program #571 is designed to prospectively evaluate the efficacy of drug-eluting stents (DES) in reducing aortocoronary saphenous vein bypass graft (SVG) failure when compared to bare metal stents (BMS) in patients undergoing stenting of de novo SVG lesions.

SVGs often develop luminal stenoses that are most commonly treated with stent implantation. Approximately 60,000-100,000 percutaneous SVG interventions are performed annually in the USA. Two types of coronary stents are currently available: bare metal stents and drug eluting stents. Bare metal stents are the standard of care for the percutaneous treatment of SVG lesions, but are limited by high rates of in-stent restenosis (as high as 51% after 12 months) often leading to repeat percutaneous or surgical SVG treatments. Drug-eluting stents have been shown to significantly reduce in-stent restenosis and the need for repeat target vessel and lesion revascularization in native coronary arteries, yet their efficacy in SVGs is not well studied, with conflicting results from various small studies. The proposed Cooperative Studies Program study will be the first large prospective, randomized, multicenter, blinded clinical trial comparing DES and BMS in SVG lesions. It will provide critical knowledge to assist the cardiac interventionalist in selecting the optimum stent type for these challenging lesions.

Patients undergoing clinically-indicated stenting of de novo SVG lesions will be randomized in a 1:1 ratio to DES or BMS. To ensure blinding to the type of stent used, of the patients who do not present with an acute coronary syndrome and do not require 12 months of dual antiplatelet therapy, those who receive DES will receive 11 months of clopidogrel and those who receive BMS will receive 11 months of matching placebo. After stenting, patients will be followed clinically for a minimum of one year to determine the 12-month incidence of target vessel failure (TVF, primary study endpoint). TVF will be defined as the composite of cardiac death, target vessel myocardial infarction and target vessel revascularization, and is the primary clinical endpoint used in all FDA-approved DES pivotal trials. Coronary angiography and intervention during follow-up will only be performed if clinically-indicated (no mandatory angiographic follow-up). Secondary endpoints include: 1) clinical outcomes other than TVF (procedural success; post-procedural myocardial infarction; post-procedural bleeding; all cause death and cardiac death; follow-up myocardial infarction; stent thrombosis; target lesion revascularization; target vessel revascularization; non-target vessel revascularization; the composite endpoint of death, myocardial infarction, and target vessel revascularization (patient-oriented composite endpoint according to the FDA guidance document on DES studies); the composite endpoint of cardiac death, target vessel myocardial infarction, and target lesion revascularization (device-oriented composite endpoint for target lesion failure); and stroke); and 2) incremental cost-effectiveness of DES relative to BMS. A tertiary endpoint is in-stent neointima proliferation as measured by intravascular ultrasonography.

Based on published studies, the investigators estimate the 12-month TVF rate in the BMS arm to be 30%. The investigators hypothesize that DES will reduce TVF to 18% (40% relative reduction). Assuming two-year accrual and one interim assessment, a total sample size of about 520 patients will be needed to detect this difference with 90% power, using a two-sided 5% significance level. Assuming an intake rate of 1 patient per month per VA Medical Center, the investigators will need 22 participating sites. However, the investigators will begin the study with 25 sites to protect against a site dropout rate of 10%.

Percutaneous treatment of SVG lesions is of particular importance to the VA system because many Veterans have undergone and continue to undergo coronary artery bypass graft surgery. Every year, approximately 12-15% of percutaneous coronary interventions performed within the VA system are performed in SVGs, at a cost of approximately $15,000-$20,000 per procedure; DES are currently used in approximately half of SVG interventions. Because of (a) the high prevalence and high cost of SVG stenting, (b) DES cost two- to three- fold more than BMS and often require prolonged ( 12 months) thienopyridine administration to prevent late stent thrombosis, and (c) DES may have increased risk for late and very late stent thrombosis, a catastrophic complication with high mortality, the proposed study will have considerable impact on the clinical practice of SVG lesion stenting, patient satisfaction, and financial burden of health care systems (both within and outside the VA), regardless of whether the results are positive (DES offer significantly superior health benefits to patients than BMS), or negative (DES do not offer significantly superior health benefits to patients than BMS). Due to decreasing profits and increasing competition, DES manufacturers are not planning to ever fund a SVG DES study. The VA system with its Cooperative Studies Program is uniquely suited to conduct the proposed study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years
* Need for percutaneous coronary intervention of a 50-99% de novo SVG lesion that is between 2.25 and 4.5 mm in diameter and that is considered to cause clinical or functional ischemia
* Intent to use a distal embolic protection device
* Agrees to participate and to take prescribed medications as instructed
* Has provided informed consent and agrees to participate

Exclusion Criteria:

* Planned non-cardiac surgery within the following 12 months
* Presentation with an ST-segment elevation acute myocardial infarction
* Target SVG is the last remaining vessel or is the "left main" equivalent
* Any previous percutaneous treatment of the target lesion (with balloon angioplasty, stent, intravascular brachytherapy etc)
* Any previous percutaneous treatment of the target vessel (of a lesion different than the target lesion) within the prior 12 months
* Hemorrhagic diatheses, or refusal to receive blood transfusions
* Warfarin administration required for the next 12 months and patient considered to be at high risk of bleeding with triple anticoagulation/antiplatelet therapy
* Recent positive pregnancy test, breast-feeding, or possibility of a future pregnancy (defined as no prior hysterectomy or as <5 years elapsing since last menstrual period)
* Coexisting conditions that limit life expectancy to less than 12 months
* History of an allergic reaction or significant sensitivity to drugs such as sirolimus, paclitaxel, zotarolimus, or everolimus included in various DES. History of an allergic reaction or significant sensitivity to L-605 cobalt chromium alloy (cobalt, silicon, chromium, tungsten, manganese, iron, nickel), F562 cobalt chromium alloy (cobalt, chromium, nickel), 316L surgical stainless steel (iron, chromium, nickel, and molybdenum), or MP35N cobalt-based alloy (cobalt, nickel, chromium, molybdenum, titanium, iron, silicon, and manganese), or components of the platinum chromium alloy stent.
* Allergy to clopidogrel in patients who do not present with an acute coronary syndrome (ACS), where ACS is defined as cardiac ischemic symptoms occurring at rest and 1 of the following 3 criteria: electrocardiographic changes suggestive of ischemia (ST-segment elevation or depression 1 mm in 2 contiguous leads, or new left bundle branch block, or posterior myocardial infarction); positive biomarker indicating myocardial necrosis (troponin I or T or creatine kinase-MB greater than the upper limit of normal); or coronary revascularization performed during hospitalization triggered by the cardiac ischemic symptoms
* Participating in another interventional randomized trial (required condition for all CSP studies) for which dual enrollment with DIVA is not approved

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 597 (Actual)
Dates: Start 2012-01-11 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanouil S Brilakis, MD PhD, Study Chair — VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX; Subhash Banerjee, MD, Study Chair — VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX
Locations (25):
- United States (25):
  - Southern Arizona VA Health Care System, Tucson, AZ, Tucson, Arizona
  - Central Arkansas VHS John L. McClellan Memorial Veterans Hospital, Little Rock, AR, Little Rock, Arkansas
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - VA Eastern Colorado Health Care System, Denver, CO, Denver, Colorado
  - Washington DC VA Medical Center, Washington, DC, Washington D.C., District of Columbia
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana
  - Lexington VA Medical Center, Lexington, KY, Lexington, Kentucky
  - Southeast Louisiana Veterans Health Care System, New Orleans, LA, New Orleans, Louisiana
  - VA Boston Healthcare System West Roxbury Campus, West Roxbury, MA, West Roxbury, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Harry S. Truman Memorial, Columbia, MO, Columbia, Missouri
  - St. Louis VA Medical Center John Cochran Division, St. Louis, MO, St Louis, Missouri
  - Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY, New York, New York
  - Asheville VA Medical Center, Asheville, NC, Asheville, North Carolina
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - Oklahoma City VA Medical Center, Oklahoma City, OK, Oklahoma City, Oklahoma
  - Memphis VA Medical Center, Memphis, TN, Memphis, Tennessee
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xenogiannis I, Rangan BV, Uyeda L, Banerjee S, Edson R, Bhatt DL, Goldman S, Holmes DR Jr, Rao SV, Shunk K, Mavromatis K, Ramanathan K, Bavry AA, McFalls EO, Garcia S, Thai H, Uretsky BF, Latif F, Armstrong E, Ortiz J, Jneid H, Liu J, Aggrawal K, Conner TA, Wagner T, Karacsonyi J, Ventura B, Alsleben A, Lu Y, Shih MC, Brilakis ES. In-Stent Restenosis in Saphenous Vein Grafts (from the DIVA Trial). Am J Cardiol. 2022 Jan 1;162:24-30. doi: 10.1016/j.amjcard.2021.09.024. Epub 2021 Nov 1. PMID 34736721
- [Derived] Latif F, Uyeda L, Edson R, Bhatt DL, Goldman S, Holmes DR Jr, Rao SV, Shunk K, Aggarwal K, Uretsky B, Bolad I, Ziada K, McFalls E, Irimpen A, Truong HT, Kinlay S, Papademetriou V, Velagaleti RS, Rangan BV, Mavromatis K, Shih MC, Banerjee S, Brilakis ES. Stent-Only Versus Adjunctive Balloon Angioplasty Approach for Saphenous Vein Graft Percutaneous Coronary Intervention: Insights From DIVA Trial. Circ Cardiovasc Interv. 2020 Feb;13(2):e008494. doi: 10.1161/CIRCINTERVENTIONS.119.008494. Epub 2020 Feb 5. PMID 32019343
- [Derived] Brilakis ES, Edson R, Bhatt DL, Goldman S, Holmes DR Jr, Rao SV, Shunk K, Rangan BV, Mavromatis K, Ramanathan K, Bavry AA, Garcia S, Latif F, Armstrong E, Jneid H, Conner TA, Wagner T, Karacsonyi J, Uyeda L, Ventura B, Alsleben A, Lu Y, Shih MC, Banerjee S; DIVA Trial Investigators. Drug-eluting stents versus bare-metal stents in saphenous vein grafts: a double-blind, randomised trial. Lancet. 2018 May 19;391(10134):1997-2007. doi: 10.1016/S0140-6736(18)30801-8. Epub 2018 May 11. PMID 29759512

RESULTS

PARTICIPANT FLOW:
Groups:
- Bare Metal Stent Group: Patients who receive a bare metal stent (BMS) in the saphenous vein graft target lesion(s).
  Bare Metal Stent: Patients receive one or more bare metal stents in the saphenous vein graft target lesion.
  Placebo: For non-acute coronary syndrome (ACS) patients with no other clinical indication for open-label thienopyridine who receive only BMS.
  Thienopyridine (open-label): For ACS patients who receive BMS or Drug Eluting Stent (DES) in their saphenous vein graft or patients for whom there is another clinical indication for open-label thienopyridine. Also for patients who receive a DES in a non-target lesion.
- Drug Eluting Stent Group: Patients who receive a drug-eluting stent (DES) in the saphenous vein graft target lesion(s).
  Drug-Eluting Stent: Patients receive one or more drug-eluting stents in the saphenous vein graft target lesion.
  Blinded clopidogrel: For non-acute coronary syndrome (ACS) patients with no other clinical indication for open-label thienopyridine who receive one or more DES in the target lesion.
  Thienopyridine (open-label): For ACS patients who receive Bare Metal Stent (BMS) or DES in their saphenous vein graft or patients for whom there is another clinical indication for open-label thienopyridine. Also for patients who receive a DES in a non-target lesion.
Period: Overall Study
Arm/Group | Bare Metal Stent Group | Drug Eluting Stent Group
Started | 305 | 292
Completed | 280 | 275
Not Completed | 25 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BMS Group | DES Group | Total
Number analyzed (Participants) | 305 | 292 | 597
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (7.7) | 69.0 (7.4) | 68.6 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 305 | 290 | 595
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 16 | 30
  Not Hispanic or Latino | 286 | 270 | 556
  Unknown or Not Reported | 5 | 6 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 254 | 263 | 517
  Black/African American | 32 | 17 | 49
  Other | 13 | 7 | 20
  Not Answered | 6 | 5 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 305 | 292 | 597

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Target Vessel Failure (TVF), Defined as the Composite of Cardiac Death
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | BMS Group | DES Group
Number analyzed (Participants) | 305 | 292
Participants | 16 | 17

2. Primary Outcome: Number of Participants With Target Vessel Failure (TVF), Defined as the Target Vessel Myocardial Infarction
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bare Metal Stent Group | Drug Eluting Stent Group
Number analyzed (Participants) | 305 | 292
Participants | 20 | 16

3. Primary Outcome: Number of Participants With Target Vessel Failure (TVF), Defined as the Target Vessel Revascularization
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bare Metal Stent Group | Drug Eluting Stent Group
Number analyzed (Participants) | 305 | 292
Participants | 34 | 34

4. Secondary Outcome: Incremental Cost-effectiveness of DES Relative to BMS
Time Frame: 12 months
Measure: Mean (Standard Error); unit: U.S. Dollars
Arm/Group | Bare Metal Stent Group | Drug Eluting Stent Group
Number analyzed (Participants) | 305 | 292
U.S. Dollars | 20939 (1051) | 21051 (1075)

5. Secondary Outcome: Procedural Success
Description: The procedural success rate and the incidence of post-procedural myocardial infarction and post-procedural GUSTO moderate or severe bleeding were compared between the DES and BMS groups by the difference between two independent proportions. Cumulative incidence curves and stratified log-rank tests were used to compare the two stent groups on the incidence of the secondary clinical outcomes listed above. When appropriate, competing risks analyses with plots of cumulative incidence curves and comparisons of cumulative incidences with Gray's test and Fine and Gray's methods were done. Proportional hazards regression for sub-distributions of competing risks were also done. SAS 9.2 (TS2M3; SAS Institute, Cary, NC, USA) and R version 3.4.4 were used for the analyses.
Time Frame: Discharge from Index Hospitalization (an average of 36 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Bare Metal Stent Group | Drug Eluting Stent Group
Number analyzed (Participants) | 305 | 292
Participants | 291 | 274

6. Secondary Outcome: Number of Participant Deaths (All Cause and Cardiac). All Deaths Will be Considered Cardiac Unless an Unequivocal Non-cardiac Cause Can be Established.
Time Frame: Entire Duration of Follow-up (median 2.7 years)
Measure: Count of Participants; unit: Participants
Arm/Group | BMS Group | DES Group
Number analyzed (Participants) | 305 | 292
Participants | 51 | 55

7. Secondary Outcome: Number of Participants With Myocardial Infarction (MI)
Time Frame: Entire Duration of Follow-up (median 2.7 years)
Measure: Count of Participants; unit: Participants
Arm/Group | BMS Group | DES Group
Number analyzed (Participants) | 305 | 292
Participants | 62 | 53

8. Secondary Outcome: Number of Participants With Definite Stent Thrombosis as Defined Using the Academic Research Consortium (ARC) Definition
Description: Definite stent thrombosis will be considered to have occurred by either angiographic or pathologic confirmation.
  Angiographic Confirmation of Stent Thrombosis will be defined as the presence of thrombus originating in a study stent, or in the segment 5mm proximal or distal to the stent AND fulfillment of at least one of the following 5 criteria within a 48 hour time window:
  * Acute onset of ischemic symptoms at rest
  * New ischemic ECG changes suggestive of acute ischemia
  * Rise and fall of cardiac biomarkers
  * Nonocclusive intracoronary thrombus seen in multiple projections, or persistence of contrast material within the lumen, or a visible embolization of intraluminal material downstream
  * Occlusive intracoronary thrombus Pathological Confirmation of stent thrombosis will be defined as evidence of recent thrombus with the stent determined at autopsy or via examination of tissue retrieved following thrombectomy.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | BMS Group | DES Group
Number analyzed (Participants) | 305 | 292
Participants | 7 | 6

9. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Time Frame: Entire Duration of Follow-up (median 2.7 years)
Measure: Count of Participants; unit: Participants
Arm/Group | BMS Group | DES Group
Number analyzed (Participants) | 305 | 292
Participants | 105 | 108

10. Secondary Outcome: Patient-Oriented Composite Endpoint Will be Used as Secondary Outcome
Description: The patient-oriented composite endpoint is defined as the composite of all-cause death, any myocardial infarction and target vessel revascularization.
  Target vessel (SVG) revascularization (TVR) will be defined as any repeat percutaneous intervention or surgical bypass of any segment of the target SVG and the native coronary vessel distal to the SVG anastomosis. Non-target vessel revascularization will be defined as any repeat percutaneous intervention or surgical bypass of any SVG or any native coronary vessel apart from the target SVG and the native coronary artery supplied by the target SVG.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bare Metal Stent Group | Drug Eluting Stent Group
Number analyzed (Participants) | 305 | 292
Participants | 68 | 62

11. Secondary Outcome: In Patients Who Clinically Require Follow-up Angiography, Two Angiographic Endpoints Will be Assessed: (a) In-segment Binary Restenosis and (b) Angiographic Late In-segment Luminal Loss.
Description: This outcome is for the in-segment binary restenosis.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bare Metal Stent Group | Drug Eluting Stent Group
Number analyzed (Participants) | 137 | 139
Participants | 57 | 56

12. Secondary Outcome: Number of Participants With Stroke
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bare Metal Stent Group | Drug Eluting Stent Group
Number analyzed (Participants) | 305 | 292
Participants | 3 | 2

13. Secondary Outcome: Incremental Cost-effectiveness Ratios (ICERs) for Subgroups of Patients, Such as Those With Highest Risk of Restenosis, Tallies of Cost by Type, and a Cost-outcomes Analysis Such as Cost Per Restenosis Avoided.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: U.S. Dollars
Groups:
- Diabetes; Number of Lesions (1 Lesion); Number of Lesions (2 or More Lesions); Stent Diameter (2.25 to Less Than 3); Stent Diameter (3 to Less Than 3.5); Stent Diameter (3.5 to Less Than 4); Recipient Target Vessel (Laddiag); Recipient Target Vessel (Cxom); Lesion Location (Aortic/Ostial); Lesion Location (Body); Antiplatelet; Baseline ACS Score: Interaction effects of this DES Subgroup
Arm/Group | Diabetes | Number of Lesions (1 Lesion) | Number of Lesions (2 or More Lesions) | Stent Diameter (2.25 to Less Than 3) | Stent Diameter (3 to Less Than 3.5) | Stent Diameter (3.5 to Less Than 4) | Recipient Target Vessel (Laddiag) | Recipient Target Vessel (Cxom) | Lesion Location (Aortic/Ostial) | Lesion Location (Body) | Antiplatelet | Baseline ACS Score
Number analyzed (Participants) | 292 | 292 | 292 | 292 | 292 | 292 | 292 | 292 | 292 | 292 | 292 | 292
U.S. Dollars | -2578.71 (3059.08) | -2971.90 (22,730.43) | -17998.43 (23914.95) | -11768.06 (4723.68) | -5069.18 (4448.96) | -14152 (4550.29) | -771.50 (4073.11) | -4,487.11 (4082.83) | 8433.33 (3598.76) | 4780.21 (5671.55) | -1483.97 (3062.72) | -3733.04 (3038.69)

14. Secondary Outcome: In-stent Neointima Proliferation as Measured by Intravascular Ultrasonography
Time Frame: 12 months
Population: The study did not collect information needed from the IVUS procedures to calculate neointima proliferation.
Arm/Group | Bare Metal Stent Group | Drug Eluting Stent Group
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | BMS Group | DES Group
Number analyzed (Participants) | 305 | 292
Participants | 25 | 26

16. Secondary Outcome: Number of Participants With Target Vessel Myocardial Infarction
Time Frame: Entire Duration of Follow-up (median 2.7 years)
Measure: Count of Participants; unit: Participants
Arm/Group | BMS Group | DES Group
Number analyzed (Participants) | 305 | 292
Participants | 40 | 35

17. Secondary Outcome: Number of Participants With Any Revascularization
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | BMS Group | DES Group
Number analyzed (Participants) | 305 | 292
Participants | 53 | 56

18. Secondary Outcome: Number of Participants With Definite or Probable Stent Thrombosis
Description: Definite stent thrombosis will be considered to have occurred by either angiographic or pathologic confirmation.
  Probable Stent Thrombosis will clinically be considered to have occurred after index Saphenous Vein aortocoronary bypass Graft (SVG) stenting (the Percutaneous Coronary Intervention (PCI) immediately after randomization) in the following cases: a) any unexplained death within the first 30 days OR b) Irrespective of the time after the index procedure, any MI which is related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation of stent thrombosis and in the absence of any other obvious cause.
Time Frame: Entire Duration of Follow-up (median 2.7 years)
Measure: Count of Participants; unit: Participants
Arm/Group | BMS Group | DES Group
Number analyzed (Participants) | 305 | 292
Participants | 30 | 26

19. Secondary Outcome: Procedural Complications (Post-procedural Myocardial Infarction and Post-procedural Bleeding)
Description: Incidence of post-procedural myocardial infarction and post-procedural GUSTO moderate or severe bleeding were compared between the DES and BMS groups by the difference between two independent proportions. Cumulative incidence curves and stratified log-rank tests were used to compare the two stent groups on the incidence of the secondary clinical outcomes listed above. When appropriate, competing risks analyses with plots of cumulative incidence curves and comparisons of cumulative incidences with Gray's test and Fine and Gray's methods were done. Proportional hazards regression for sub-distributions of competing risks were also done. SAS 9.2 (TS2M3; SAS Institute, Cary, NC, USA) and R version 3.4.4 were used for the analyses.
Time Frame: Discharge from Index Hospitalization (an average of 36 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Bare Metal Stent Group | Drug Eluting Stent Group
Number analyzed (Participants) | 305 | 292
Participants | 22 | 15

20. Secondary Outcome: Device-oriented Composite Endpoint of Target Lesion Failure Will be Used as a Secondary Outcome
Description: The Device-oriented composite endpoint of Target lesion failure is defined as the composite of cardiac or unknown death, target vessel myocardial infarction, and target lesion revascularization.
  Target lesion revascularization (TLR) will be defined as any repeat percutaneous intervention of the target SVG lesion or bypass surgery of the target SVG lesion performed for restenosis or other complication of the target lesion. The target lesion will be defined as the treated SVG segment from 5 mm proximal to the stent to 5 mm distal to the stent.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bare Metal Stent Group | Drug Eluting Stent Group
Number analyzed (Participants) | 305 | 292
Participants | 51 | 45

21. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Time Frame: Entire Duration of Follow-up (median 2.7 years)
Measure: Count of Participants; unit: Participants
Arm/Group | BMS Group | DES Group
Number analyzed (Participants) | 305 | 292
Participants | 40 | 47

22. Secondary Outcome: Number of Participants With Non-Target Revascularization
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bare Metal Stent Group | Drug Eluting Stent Group
Number analyzed (Participants) | 305 | 292
Participants | 26 | 33

23. Secondary Outcome: Number of Participants With Non-Target Revascularization
Time Frame: Entire Duration of Follow-up (median 2.7 years)
Measure: Count of Participants; unit: Participants
Arm/Group | Bare Metal Stent Group | Drug Eluting Stent Group
Number analyzed (Participants) | 305 | 292
Participants | 60 | 69

24. Secondary Outcome: Patient-oriented (for Target Lesion Failure) Composite Endpoints Will be Used as Secondary Outcomes as Proposed by Cutlip et al, and as Recommended in the Draft FDA Guidance for Industry Statement.
Description: The patient-oriented composite endpoint is defined as the composite endpoint of any death, any myocardial infarction, or target vessel revascularization.
Time Frame: Entire Duration of Follow-up (median 2.7 years)
Measure: Count of Participants; unit: Participants
Arm/Group | Bare Metal Stent Group | Drug Eluting Stent Group
Number analyzed (Participants) | 305 | 292
Participants | 127 | 127

25. Secondary Outcome: Device-oriented (for Target Lesion Failure) Composite Endpoints Will be Used as Secondary Outcomes as Proposed by Cutlip et al, and as Recommended in the Draft FDA Guidance for Industry Statement.
Description: The device-oriented composite endpoint for target lesion failure is defined as the composite endpoint of cardiac death, target vessel myocardial infarction, or target lesion revascularization.
Time Frame: Entire Duration of Follow-up (median 2.7 years)
Measure: Count of Participants; unit: Participants
Arm/Group | Bare Metal Stent Group | Drug Eluting Stent Group
Number analyzed (Participants) | 305 | 292
Participants | 95 | 94

26. Secondary Outcome: Number of Participants With Stroke
Time Frame: Entire Duration of Follow-up (median 2.7 years)
Measure: Count of Participants; unit: Participants
Arm/Group | Bare Metal Stent Group | Drug Eluting Stent Group
Number analyzed (Participants) | 305 | 292
Participants | 12 | 10

27. Secondary Outcome: Quality Adjusted Life Years of DES Relative to BMS
Time Frame: 12 months
Measure: Mean (Standard Error); unit: years
Arm/Group | Bare Metal Stent Group | Drug Eluting Stent Group
Number analyzed (Participants) | 305 | 292
years | 0.467 (0.017) | 0.503 (0.018)

28. Secondary Outcome: Quality Adjusted Life Years for Subgroups of Patients
Time Frame: 12 months
Measure: Mean (Standard Error); unit: years
Arm/Group | Diabetes | Number of Lesions (1 Lesion) | Number of Lesions (2 or More Lesions) | Stent Diameter (2.25 to Less Than 3) | Stent Diameter (3 to Less Than 3.5) | Stent Diameter (3.5 to Less Than 4) | Recipient Target Vessel (Laddiag) | Recipient Target Vessel (Cxom) | Lesion Location (Aortic/Ostial) | Lesion Location (Body) | Antiplatelet | Baseline ACS Score
Number analyzed (Participants) | 292 | 292 | 292 | 292 | 292 | 292 | 292 | 292 | 292 | 292 | 292 | 292
years | -0.03 (0.05) | -0.04 (0.21) | -0.03 (0.19) | 0.03 (0.08) | 0.02 (0.07) | 0.04 (0.07) | -0.04 (0.07) | -0.13 (0.07) | -0.15 (0.06) | 0.02 (0.09) | -0.04 (0.05) | -0.01 (0.05)

29. Secondary Outcome: In Patients Who Clinically Require Follow-up Angiography, Two Angiographic Endpoints Will be Assessed: (a) In-segment Binary Restenosis and (b) Angiographic Late In-segment Luminal Loss.
Description: This outcome is for the angiographic late in-segment luminal loss.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Bare Metal Stent Group | Drug Eluting Stent Group
Number analyzed (Participants) | 137 | 139
lesions | 1.05 (1.21) | 0.96 (1.15)

ADVERSE EVENTS:
Time Frame: Active monitoring of Adverse Events (AEs) started once a participant is randomized at the following time periods: 18-24 hours post procedure, hospital discharge, 1 month, 3 month, 6 month, 9 month, 12 month, 18 month, 24 month, 30 month and end of study (after 12-60 months of follow-up depending on when the patient was randomized during the enrollment period).
Arm/Group | BMS Group | DES Group
All-Cause Mortality (participants affected / at risk) | 58/305 | 57/292
Serious Adverse Events (participants affected / at risk) | 244/305 | 231/292
Other Adverse Events (participants affected / at risk) | 18/305 | 12/292
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMS Group (N=305) | DES Group (N=292)
ACS/MI (Cardiac disorders) | 100 (166) | 92 (142)
Stroke (Cardiac disorders) | 17 (18) | 14 (18)
Bleed (Cardiac disorders) | 29 (41) | 28 (36)
Stent Thrombosis (Cardiac disorders) | 17 (18) | 11 (11)
Other (Cardiac disorders) | 219 (866) | 216 (859)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMS Group (N=305) | DES Group (N=292)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (6)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes